CLINICAL TRIAL: NCT02264496
Title: The Effects of Exercise on Outcomes in Patients Undergoing Surgery for Colorectal Cancer: a Pilot Prospective Randomised Trial.
Brief Title: Prospective Randomised Trial of Exercise and / or Antioxidants in COlorectal Cancer Patients Undergoing Surgery.
Acronym: PEACOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/YH/0322 V3
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Exercise; CPEX; Exercise, Physical; Exercise, Aerobic; Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard pre-operative care
- Exercise (Experimental): A 2-4 week low volume, moderate intensity, supervised, one to one, individualised exercise programme. '
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise

SUMMARY:
Colorectal cancer is the fourth most common cancer in the UK. Surgical resection is the mainstay of curative therapy. With the screening program enabling early detection, surgery plays an important role in treatment strategies. Surgery imparts a significant physiological and psychological stress on cancer patients.Recent research has demonstrated that a fast-track approach utilising regional anaesthesia, early mobilisation and good oral intake can improve outcomes by reducing the physiological stress response to surgery. The primary objective of this study is to determine whether a defined exercise programme can improve recovery and reduce complications after surgery.

DETAILED DESCRIPTION:
Study Design

This will be a prospective and randomised pilot clinical trial. For purposes of pragmatism, subjects and investigators will not be blinded to treatment allocation. The study is not blinded because it is impossible to blind investigators or patients to the exercise programme.

Patients undergoing major resectional surgery for colorectal cancer will be recruited from the Academic Surgical unit (ASU), Castle Hill Hospital. In total, 60 participants will be recruited for this pilot study and randomly allocated into 2 groups as outlined below.

The study will necessitate all participants being involved in a baseline assessment which will take on average 60 minutes with patients attending Castle Hill Hospital. Travel costs will be met.

All participants will be asked for a 15 ml blood samples on entry into the study and at 24-48 hrs prior to surgery. Regardless of recruitment, blood samples are necessary for clinical purposes at these stages in all patients as part of routine preoperative assessment prior to colorectal surgery. The aim of this is to permit an analysis of possible changes in antioxidant status prior to surgery but after preconditioning. This would be in addition to routine blood samples required.

The two groups in this study are described in more detail below. Both groups shall receive the same standard care as is normal for patients undergoing colorectal resection surgery. The only difference between groups shall be the addition of exercise preconditioning sessions to group 1. We anticipate that these will be three times a week and lasting of 60-90 minutes duration each. Travel costs will be met.

Groups

The 60 patients in this study will be randomised to one of two groups as follows:

* Group 1 - Standard care + Exercise intervention. Patients in this group will participate in a 2-4 week low volume, moderate intensity, supervised, one to one, individualised exercise programme.
* Group 2 - Standard care (Control) group. These patients will not be entered into a supervised exercise programme.

Research hypothesis 1

H0 - A two to four week period of low to moderate intensity exercise prior to surgery using an individualised exercise intervention will not reduce post-surgical length of hospital stay in colorectal cancer patients.

H1- A two to four week period of low to moderate intensity exercise prior to surgery using an individualised exercise intervention will reduce post-surgical length of hospital stay in colorectal cancer patients.

Research hypothesis 2

H0 - A two to four week period of low to moderate intensity exercise prior to surgery using an individualised exercise intervention will not modify the body's defence systems against a future oxidative stress.

H1- A two to four week period of low to moderate intensity exercise prior to surgery using an individualised exercise intervention will modify the body's defence systems against a future oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with colorectal cancer listed for elective resection surgery who have consented to participate in the study.

Exclusion Criteria:

* History of unstable angina/unstable coronary artery disease or a heart attack in the previous month
* Any heart related disease including but not limited to aortic stenosis, pericarditis or any thromboembolic disease
* Severe Infections and fever
* Uncontrolled metabolic diseases
* Uncontrolled asthma
* Acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
* Resting heart rate of more than 120 BPM
* Systolic blood pressure of more than 180 mm Hg or diastolic blood pressure of more than 110 mm Hg
* Recent cerebrovascular accident
* Pregnancy
* Preexisting severe physical disability
* Age <18 years
* Unwilling to allow their GP to be informed of their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Length of stay | Up to 3 months
  Post-operative hospital length of stay until medically fit for discharge.

SECONDARY OUTCOMES:
Antioxidant capacity | Up to 4 weeks
  Biochemical markers of antioxidant capacity: Hsp 32/72, CD11b/CD18 and Glutathione measured pre- and post-intervention.
Exercise capacity | Up to 3 months
  Exercise test and CPEX parameters assessed pre-intervention, post-intervention and at 3 months post surgery.
Complications | Up to 3 months
  All post-operative complications assessed at 3 months post surgery.
Quality of Life Questionnaires | Up to 3 months
  Validated QOL questionnaires completed pre-intervention, post-intervention and at 3 months post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John Hartley, MD FRCS, Principal Investigator — Hull and East Yorkshire NHS Trust
Locations (1):
- Academic Surgical Unit, Castle Hill Hospital, Hull, East Yorkshire, United Kingdom